CLINICAL TRIAL: NCT02626845
Title: Rituximab for the Otolaryngologic Manifestations of Granulomatosis With Polyangiitis
Acronym: RENTGPA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Genentech, Inc. (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-424
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Granulomatosis With Polyangiitis (Wegener's Granulomatosis)
Keywords: Granulomatosis with Polyangiitis; Wegener's Granulomatosis; GPA; Rituximab; Rituxan; ENT GPA
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab Arm (Active Comparator): All subjects in this arm will receive standard of care induction therapy, and then will receive two additional rituximab infusions at week 16 and week 32.
  Interventions: Drug: Rituximab
- Placebo Arm (Placebo Comparator): All subjects in this arm will receive standard of care induction therapy, and then will receive two additional placebo infusions at week 16 and week 32.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rituximab — Standard of care induction with Rituximab: 375mg/m2 weekly x 4 weeks. Once randomized, the rituximab dose will be 1000mg IV every 4 months x 2.
  Other Names: Rituxan
  Arms: Rituximab Arm
Other: Placebo — Will be given at two time-points (week 16 and week 32) to subjects in the Placebo Arm.
  Arms: Placebo Arm

SUMMARY:
This is a phase IV, single-center, randomized, placebo-controlled pilot study that will evaluate the efficacy of rituximab at inducing otolaryngologic remission in GPA patients with active otolaryngologic disease.

DETAILED DESCRIPTION:
Patients with GPA and active ENT disease in at least two ENT domains, as defined after endoscopic visualization of the upper airway and audiometric evaluation by a single otolaryngologist using a validated GPA ENT disease activity score, will be eligible for inclusion. ENT disease may be new, grumbling or relapsing.

All patients entering the trial will receive standard induction therapy with rituximab (375mg/m2 per week x 4). At week 16, patients will be randomized to receive maintenance rituximab (1000mg) every 4 months or placebo infusions. The primary outcome will be assessed at week 52. Patients will be treated with a standardized prednisone taper according to whether they had severe or limited disease at study entry, prednisone taper will be completed at week 16.

The investigators plan to enroll 28 patients who will be randomized in a 1:1 fashion to rituximab or placebo. The investigators estimate accrual of these subjects will take 18 months from study initiation. Once enrolled, subjects are followed for 52 weeks until the primary endpoint is assessed.

ELIGIBILITY:
Inclusion Criteria:

GPA Specific Inclusion:

1. Patients must have met at least 2 of the 5 modified ACR classification criteria for GPA. These do not need to be present at the time of study entry. The modified ACR criteria are:

   * Nasal or oral inflammation, defined as the development of painful or painless oral ulcers or purulent or bloody nasal discharge
   * Abnormal chest radiograph, defined as the presence of nodules, fixed infiltrates, or cavities
   * Active urinary sediment, defined as microscopic hematuria (>5 red blood cells per high power field) or red blood cell casts
   * Granulomatous inflammation on biopsy, defined as histologic changes showing granulomatous inflammation within the wall of an artery or in the perivascular or extravascular area (artery or arteriole)
   * Positive anti-neutrophil cytoplasmic antibody (ANCA) test specific for proteinase-3, measured by enzyme-linked immunoassay
2. Active GPA in the ENT domain within 1 month prior to screening, where the active disease is defined as a score of ≥2 on a GPA ENT disease activity score (7 items scored as 1= present 0= absent) performed by direct endoscopic visualization of the upper airway and audiometric evaluation by a single expert otolaryngologist. Items included in the GPA ENT disease activity score are:

   * Bloody rhinorrhea (Daily blood stained nasal discharge)
   * Objective stridor (Stridor assessed by doctor)
   * Inflammation on nasal examination (Ulcers, granulation, friable mucosa on rigid nasendoscopy. Excluding crusting)
   * Inflammation on flexible laryngoscopy (Ulcers, granulation, friable mucosa in the larynx)
   * Inflamed TM*/middle ear (Persistent inflammation or granulation tissue in tympanic membrane/middle ear)
   * Sudden sensorineural hearing loss (30db drop in 3 frequencies within 72 hours)
   * Other ENT/upper airway manifestations of active GPA observed during structured ENT exam including but not limited to lacrimal gland dacryocystitis and endobronchial disease

   General Medical Concerns:
3. Age 18 and older
4. Willing and able to comply with treatment and follow-up procedures
5. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment.
6. Willing and able to provide written informed consent

Rituximab-Specific Concerns:

* ANC: > 1000/mm3
* Platelets: > 100,000/mm3
* Hemoglobin: > 7 gm/dL
* Adequate renal function as indicated by Cr >4.0mg/dl
* Adequate liver function as defined by AST or ALT <2x Upper Limit of Normal unless related to primary disease.

Exclusion Criteria:

Disease-Specific Concerns:

1. Creatinine >4.0mg/dl
2. Respiratory failure requiring mechanical ventilatory support
3. Previous treatment with rituximab (Rituxan® ) within 6 months of screening
4. History of severe allergic or anaphylactic reaction or serious infusion reaction while receiving rituximab
5. Failure to respond to previous course of rituximab (Rituxan®) administered for treatment of GPA, as determined by the discretion of the PI

5. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies 6. Use of the maintenance immunosuppressive agent (methotrexate, azathioprine, mycophenolate mofetil or leflunomide) within 5 drug half-lives prior to baseline 7. Treatment with any other biologic agent, including belimumab, within the past 3 months of screening 8. Treatment with cyclophosphamide (oral or intravenous) within the past 1 month of screening

General Medical Concerns:

* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment), or lactating.
* Inability to comply with study and/or follow-up procedures.

Rituximab-Specific Concerns:

* History of HIV.
* Presence of active infection..
* New York Heart Association Classification III or IV heart disease (See Appendix D).
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of psychiatric disorder.
* At the Investigator's discretion, receipt of a live vaccine within 4 weeks prior to randomization.

Positive hepatitis B or C serology is considered a potential exclusion criterion. Hepatitis B screening should include hepatitis B surface antigen (HBsAg) and core antibody (anti-HBc) in all patients. For patients who show evidence of prior hepatitis B infection (HBsAg positive [regardless of antibody status] or HBsAg negative but anti-HBc positive), consult with physicians with expertise in managing hepatitis B regarding monitoring and consideration for HBV antiviral therapy before and/or during Rituxan treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in ENT remission without relapse at week 52 in each treatment group. | Assessed at week 52
  ENT remission is defined as a GPA ENT disease activity score of 0.

SECONDARY OUTCOMES:
Comparison of mean ENT disease activity scores between treatment arms | Assessed at week 52
Cumulative steroid dose | Assessed at week 52
Duration of steroid free remission | Assessed at week 52
Proportion of subject in remission without relapse and completed steroid taper | Assessed at week 52
Quality of Life as measured by the SNOT-22 Questionnaire | Assessed at week 0, 16, and 52
Change in VDI in the ENT domain | Assessed at week 52
Number of surgical procedures in the ENT domain required during the study period | Assessed at week 52
Number of ENT flares as measured by the ENT GPA DAS | Assessed at week 52
Number of GPA flares as measured by BVAS-WG | Assessed at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seo P, Min YI, Holbrook JT, Hoffman GS, Merkel PA, Spiera R, Davis JC, Ytterberg SR, St Clair EW, McCune WJ, Specks U, Allen NB, Luqmani RA, Stone JH; WGET Research Group. Damage caused by Wegener's granulomatosis and its treatment: prospective data from the Wegener's Granulomatosis Etanercept Trial (WGET). Arthritis Rheum. 2005 Jul;52(7):2168-78. doi: 10.1002/art.21117. PMID 15986348
- [Background] Hogan SL, Falk RJ, Chin H, Cai J, Jennette CE, Jennette JC, Nachman PH. Predictors of relapse and treatment resistance in antineutrophil cytoplasmic antibody-associated small-vessel vasculitis. Ann Intern Med. 2005 Nov 1;143(9):621-31. doi: 10.7326/0003-4819-143-9-200511010-00005. PMID 16263884
- [Background] Srouji IA, Andrews P, Edwards C, Lund VJ. General and rhinosinusitis-related quality of life in patients with Wegener's granulomatosis. Laryngoscope. 2006 Sep;116(9):1621-5. doi: 10.1097/01.mlg.0000230440.83375.4b. PMID 16954992
- [Background] Hoffman GS, Kerr GS, Leavitt RY, Hallahan CW, Lebovics RS, Travis WD, Rottem M, Fauci AS. Wegener granulomatosis: an analysis of 158 patients. Ann Intern Med. 1992 Mar 15;116(6):488-98. doi: 10.7326/0003-4819-116-6-488. PMID 1739240
- [Background] Stone JH; Wegener's Granulomatosis Etanercept Trial Research Group. Limited versus severe Wegener's granulomatosis: baseline data on patients in the Wegener's granulomatosis etanercept trial. Arthritis Rheum. 2003 Aug;48(8):2299-309. doi: 10.1002/art.11075. PMID 12905485
- [Background] De Groot K, Rasmussen N, Bacon PA, Tervaert JW, Feighery C, Gregorini G, Gross WL, Luqmani R, Jayne DR. Randomized trial of cyclophosphamide versus methotrexate for induction of remission in early systemic antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2005 Aug;52(8):2461-9. doi: 10.1002/art.21142. PMID 16052573
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Jones RB, Furuta S, Tervaert JW, Hauser T, Luqmani R, Morgan MD, Peh CA, Savage CO, Segelmark M, Tesar V, van Paassen P, Walsh M, Westman K, Jayne DR; European Vasculitis Society (EUVAS). Rituximab versus cyclophosphamide in ANCA-associated renal vasculitis: 2-year results of a randomised trial. Ann Rheum Dis. 2015 Jun;74(6):1178-82. doi: 10.1136/annrheumdis-2014-206404. Epub 2015 Mar 4. PMID 25739829
- [Background] Specks U, Merkel PA, Seo P, Spiera R, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Fessler BJ, Ding L, Viviano L, Tchao NK, Phippard DJ, Asare AL, Lim N, Ikle D, Jepson B, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh K, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Mueller M, Sejismundo LP, Mieras K, Stone JH; RAVE-ITN Research Group. Efficacy of remission-induction regimens for ANCA-associated vasculitis. N Engl J Med. 2013 Aug 1;369(5):417-27. doi: 10.1056/NEJMoa1213277. PMID 23902481
- [Background] Aries PM, Hellmich B, Voswinkel J, Both M, Nolle B, Holl-Ulrich K, Lamprecht P, Gross WL. Lack of efficacy of rituximab in Wegener's granulomatosis with refractory granulomatous manifestations. Ann Rheum Dis. 2006 Jul;65(7):853-8. doi: 10.1136/ard.2005.044420. Epub 2005 Nov 3. PMID 16269425
- [Background] Seo P, Specks U, Keogh KA. Efficacy of rituximab in limited Wegener's granulomatosis with refractory granulomatous manifestations. J Rheumatol. 2008 Oct;35(10):2017-23. Epub 2008 Aug 1. PMID 18688911
- [Background] Martinez Del Pero M, Chaudhry A, Jones RB, Sivasothy P, Jani P, Jayne D. B-cell depletion with rituximab for refractory head and neck Wegener's granulomatosis: a cohort study. Clin Otolaryngol. 2009 Aug;34(4):328-35. doi: 10.1111/j.1749-4486.2009.01968.x. PMID 19673980
- [Background] Lally L, Lebovics RS, Huang WT, Spiera RF. Effectiveness of rituximab for the otolaryngologic manifestations of granulomatosis with polyangiitis (Wegener's). Arthritis Care Res (Hoboken). 2014 Sep;66(9):1403-9. doi: 10.1002/acr.22311. PMID 25299002
- [Background] Zhao Y, Odell E, Choong LM, Barone F, Fields P, Wilkins B, Tungekar FM, Patel P, Sanderson JD, Sangle S, D'Cruz D, Spencer J. Granulomatosis with polyangiitis involves sustained mucosal inflammation that is rich in B-cell survival factors and autoantigen. Rheumatology (Oxford). 2012 Sep;51(9):1580-6. doi: 10.1093/rheumatology/kes123. Epub 2012 May 23. PMID 22627727
- [Background] Voswinkel J, Mueller A, Kraemer JA, Lamprecht P, Herlyn K, Holl-Ulrich K, Feller AC, Pitann S, Gause A, Gross WL. B lymphocyte maturation in Wegener's granulomatosis: a comparative analysis of VH genes from endonasal lesions. Ann Rheum Dis. 2006 Jul;65(7):859-64. doi: 10.1136/ard.2005.044909. Epub 2005 Nov 16. PMID 16291812
- [Background] Thurner L, Muller A, Cerutti M, Martin T, Pasquali JL, Gross WL, Preuss KD, Pfreundschuh M, Voswinkel J. Wegener's granuloma harbors B lymphocytes with specificities against a proinflammatory transmembrane protein and a tetraspanin. J Autoimmun. 2011 Feb;36(1):87-90. doi: 10.1016/j.jaut.2010.09.002. Epub 2010 Oct 14. PMID 20951001